CLINICAL TRIAL: NCT02326610
Title: Early hGH Treatment of Symmetrically Born Small for Gestational Age Infants to Prevent Irreversible Neurologic and Psychological Damage and Sequelae
Brief Title: Early hGH Treatment of SGA Infants to Prevent Irreversible Neurologic and Psychological Damage and Sequelae
Acronym: hGH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-14-DM-0713-12-TLV
Record Dates: First submitted 2014-11-26; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Infant, Small for Gestational Age; Growth Hormone Treatment; Infant, Premature, Diseases
Keywords: Small for gestational age (SGA); Human growth hormone (hGH)
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hGH, ZOMACTON® (somatropin) (Active Comparator): For infants in the treatment group receiving ZOMACTON® (somatropin) growth hormone by injection
  Interventions: Drug: Human growth hormone,ZOMACTON® (somatropin)
- No human growth hormone (No Intervention): No growth hormone is given.

INTERVENTIONS:
Drug: Human growth hormone,ZOMACTON® (somatropin) — The initial dose will be 30µg/kg/day. The maximal dose will be 40µg/kg/day. The dose will be adjusted by monitoring the serum IGF-I level. Growth hormone will be delivered by injection.
  Arms: hGH, ZOMACTON® (somatropin)

SUMMARY:
SGA Infants who do not show a developmental catch-up growth within the first 6 months of life fall in the category of SGA children shown to have defects in the GH/IGF-I axis, resulting in partial hGH/IGF-I deficiency.

Up to 1/4 of children born SGA have neurodevelopmental deficits. The partial hGH/IGF-I deficiency in SGA children can be the major or contributory cause of to their neurodevelopmental deficits

To assess the effect of early growth hormone treatment given to symmetrical small for gestational age (SGA) infants not demonstrating catch-up growth on neurodevelopment and growth between birth and 6-12 months.

The study is an innovative research not previously performed for improving neurodevelopmental outcome of SGA infants. As this is the first study of its kind, the safety of use of GH has not been reported, however based on multiple studies assessing use of GH in infants and young children, it is reasonable to similarly expect no short and long-term adverse effects.

The study will take place at the Tel Aviv Medical Center only.

ELIGIBILITY:
Inclusion Criteria:

* Symmetrical small for gestational age at birth: weight + length+ head circumference below -2 SD for gestational age.
* Birth weight of 1200-2200 gr
* Follow-up of growth until age of 6-12 months
* Growth parameters below -2 SD at age of 6-12 months and absence of sufficient catch-up.
* Low growth hormone levels.

Exclusion Criteria:

* Chromosomal aberration
* Any congenital syndrome and any syndrome that shows a tendency to uncontrolled cell growth and to develop tumors
* Major congenital malformation (affecting growth or development)
* Congenital infection
* Exposure to teratogenic drugs or drugs affecting development during pregnancy
* Maternal drug or alcohol abuse.
* Maternal cancer as well as cancer in 1st degree relatives.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Cognitive assessments (using the Bayley Scales of Infant Development (BSID-III) | Before treatment and 1 year later
  using the Bayley Scales of Infant Development (BSID-III)
Changes in Neurological status (formal neurological examination) | Before treatment and 1 year later
  using formal neurological examination

SECONDARY OUTCOMES:
Changes in X-ray of the hand and wrist | Before treatment and 1 year later
Pediatric Quality of life Inventory: the PedsQL measure | after 1 year of treatment
Achenbach Child Behavior Checklist (CBCL) | at the end of study after 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mandel, MD, Principal Investigator — Department of Neonatology, Tel Aviv Medical Center, 64239 Tel Aviv, Israel